CLINICAL TRIAL: NCT05610020
Title: Heparin Binding Protein as a Reliable Prognostic Biomarker for Severity of Sepsis in the Intensive Care Unit
Brief Title: Heparin Binding Protein as a Prognostic Biomarker of Sepsis Severity
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Omar Hamdy, Specialist intensive care medicine, Ain Shams University
Other Study IDs: FMASU M D 159/ 2021
Record Dates: First submitted 2022-10-20; First posted 2022-11-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Sepsis; HBP
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum blood sample
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
the aim of the study is to correlate between the severity of sepsis and serum heparin binding protein in the patients admitted to ICU with sepsis., and detect its value as a prognostic biomarker in sepsis

ELIGIBILITY:
Inclusion Criteria:

* adult whose age between 20 to70 years old
* patients suffered from sepsis or septic shock (under the third international consensus definition of sepsis and septic shock)

Exclusion Criteria:

* Any pregnancy female
* Any patient who is Neutropenic secondary to malignancy
* Patients who is taking immunosuppressive therapy
* Patients who is suffering fromHematological malignancy

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult confirmed septic patients
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Evaluate the level of Heparin binding protein in relation to patient clinical improvement measured by SOFA Score | 72 hours after meeting sepsis ceriteria
  Correlates the change of the level of Heparin binding protein in ng/ml to the clinical improvement of the patients which is measured by SOFA score

SECONDARY OUTCOMES:
Heparin binding protein and mortality | 28 days after meeting sepsis ceriteria
  Correlates the change of the level of Heparin binding protein in ng/ml And how can it is used to predict mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Omar Hamdy, Minya, Egypt